CLINICAL TRIAL: NCT02204826
Title: Effects of Korean Red Ginseng on Semen Parameters in Male Infertility Patients: a Randomized, Placebo-controlled, Double-blind Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jun Park, Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRG-infertility
Record Dates: First submitted 2014-04-24; First posted 2014-07-30 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Male Infertility
Keywords: Effects of Korean Red Ginseng on semen parameters in male infertility patients: a randomized, placebo-controlled, double-blind clinical study
MeSH Terms: conditions — Infertility, Male | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- V + KRG group (n = 20) (Experimental): three capsules of KRG (500 mg/dose) daily and varicocelectomy.
  Interventions: Drug: Korean Red Ginseng (KRG); Procedure: Varicocelectomy
- non-V + KRG group (Active Comparator): three capsules of KRG (500 mg/dose) daily
  Interventions: Drug: Korean Red Ginseng (KRG)
- V + P group (n = 20) (Active Comparator): placebo capsules and varicocelectomy
  Interventions: Procedure: Varicocelectomy
- non-V + P group (Placebo Comparator): non-V + P group (n = 20) placebo capsules
  Interventions: Drug: Korean Red Ginseng (KRG)

INTERVENTIONS:
Drug: Korean Red Ginseng (KRG) — The KRG capsules were provided by Korean Ginseng Corporation (Daejeon, Korea). KRG powder was manufactured from roots of a 6-year-old red ginseng, Panax ginseng Meyer, harvested in Republic of Korea. KRG was made by steaming fresh ginseng at 90-100 ◦C for 3 h and then drying at 50-80 ◦C.
  KRG powder prepared from grinded red ginseng (KRG capsule : 500mg/capsule). KRG was analyzed by high-performance liquid chromatography. KRG extract contained major ginsenoside-Rb1: 4.26mg/g, -Rb2: 1.62mg/g, -Rc: 1.80mg/g, -Rd: 0.29mg/g, -Re: 1.71mg/g, -Rf: 0.67mg/g, -Rg1: 2.61mg/g, -Rg2: 0.20mg/g, -Rg3: 0.13mg/g, and other minor ginsenosides. During the study period, three capsules were taken daily for 12 weeks.
  Arms: V + KRG group (n = 20); non-V + KRG group; non-V + P group
Procedure: Varicocelectomy — Surgical microscope-assisted varicocelectomy using the subinguinal approach was conducted by a single surgeon.
  Arms: V + KRG group (n = 20); V + P group (n = 20)

SUMMARY:
Korean Red ginseng (KRG) has long been applied to various diseases as a health-promoting herbal medicine in Korea. Many clinical studies of ginseng have been performed to elucidate its therapeutic characteristics. KRG has been shown to be effective in many diseases, such as cancers, hypertension, Alzheimer's disease, diabetes, acquired immune deficiency syndrome, and sexual dysfunction. Several studies have indicated effects of ginseng on improving spermatogenesis in animals. The major mechanisms behind these effects were speculated to be anti-oxidant and anti-aging effects, as well as modulation of the hypothalamus-pituitary-testis axis [7 - 10]. However, there have been no controlled human clinical trials to evaluate the effects of KRG on spermatogenesis in patients with male infertility.

Only a small proportion of causes of male infertility are currently curable, including male hypogonadal disorders that can be cured by gonadotropic agents, and obstructive azoospermia that can be corrected by surgery. In addition, evidence-based medicine has revealed that most empirical treatments are ineffective. Similarly, the efficacies of carnitine, anti-estrogens, kallikrein, vitamins C and E, and glutathione have not been confirmed.

Therefore, the investigators investigated the effects of KRG on semen parameters in male infertility patients. This is the first placebo-controlled trial to evaluate the therapeutic effects of KRG in male patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be males, 25 - 45 years of age, who had complained of infertility for at least 12 months, and had no history of surgical or medical treatments for infertility.
* Increased retrograde flow in the internal spermatic vein with venous diameter > 3 mm during the Valsalva maneuver on scrotal ultrasonography was used as an indicator of varicocele [13].
* Varicocele was graded according to the criteria presented by Lyon et al. [14]: *Grade I, palpable only with the Valsalva maneuver

  * Grade II, palpable without the Valsalva maneuver
  * Grade III, visible from a distance.

Exclusion Criteria:

* A history of vasectomy or obstructive azoospermia
* Chromosomal abnormalities
* Hypogonadism or pituitary abnormalities
* Anatomical abnormality of the genitals
* Significant hepatopathy (liver enzymes elevated 2 - 3-fold higher than the normal range)
* Renal insufficiency (serum creatinine level > 2.5 mg/dL)
* Medical treatment for infertility during the past 4 weeks.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Semen parmaters change from baseline to post-treatment | Before treatment, After 14 weeks (12 week treatment and 2 week wash out periond)
  1) sperm concentration, 2) percent motility, 3) sperm viability, and 4) Kruger/strict morphology using World Health Organization (WHO) methodologies (4th edition).

SECONDARY OUTCOMES:
Changes in hormonal parameters after treatment | Before treatment, After 14 weeks (12 week treatment and 2 week wash out periond)
  Serum concentrations of FSH and LH were measured using chemiluminescence assays, and serum total testosterone was quantified by radioimmunoassay. The hormonal status of all patients was recorded at the initial screening visit and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jun Park, PhD, MD, Principal Investigator — Department of Urology, Pusan National University Hospital
Locations (1):
- Department of Urology, Pusan National University Hospital, Busan, South Korea